CLINICAL TRIAL: NCT03694119
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Positive-Controlled Study to Evaluate the Effect of Ozanimod on Pressor Response to Oral Tyramine in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Ozanimod With Tyramine to Evaluate the Effect on Pressor Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RPC01-1913; U1111-1218-6630 (Registry Identifier: WHO)
Record Dates: First submitted 2018-08-30; First posted 2018-10-03 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Ozanimod; Oral Tyramine
MeSH Terms: interventions — Phenelzine; Tyramine; ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phenelzine (Active Comparator): Following tyramine challenging in Period 1, eligible subjects randomly assigned to Phenelzine arm are receiving Phenelzine placebo BID plus ozanimod placebo QD from Days 11 to 31, then receiving Phenelzine 15mg BID plus ozanimod placebo QD from Days 32 to 38. Subjects receive second tyramine challenge from Day 39 to up to Day 49
  Interventions: Drug: Phenelzine; Drug: Tyramine; Drug: Phenelzine placebo; Drug: ozanimod placebo
- Placebo (Placebo Comparator): Following tyramine challenging in Period 1, eligible subjects randomly assigned to Placebo arm are receiving Phenelzine placebo BID plus ozanimod placebo QD from Days 11 to 38. Subjects receive second tyramine challenge from Day 39 to up to Day 49
  Interventions: Drug: Tyramine; Drug: Phenelzine placebo; Drug: ozanimod placebo
- ozanimod (Experimental): Following tyramine challenging in Period 1, eligible subjects randomly assigned to ozanimod arm are receiving Phenelzine placebo BID plus ozanimod 1.84mg QD from Days 11 to 38, including dose escalation days. Subjects receive second tyramine challenge from Day 39 to up to Day 49
  Interventions: Drug: Tyramine; Drug: Phenelzine placebo; Drug: ozanimod

INTERVENTIONS:
Drug: Phenelzine — Phenelzine
  Arms: Phenelzine
Drug: Tyramine — Tyramine
Drug: Phenelzine placebo — Phenelzine placebo
Drug: ozanimod placebo — ozanimod placebo
  Arms: Phenelzine; Placebo
Drug: ozanimod — ozanimod
  Arms: ozanimod

SUMMARY:
The purpose of this study is to evaluate the potential effect of ozanimod on pressor response when co-administered with oral tyramine in healthy adult subjects.

Study Design This is a Phase 1, randomized, double-blind (subjects and study site personnel [except pharmacist or designee] are blinded to the treatments until 7 ± 2 days postdose follow-up), placebo- and positive-controlled study.

Study design is described below:

Subjects will be screened for participation in this study within 28 days prior to dosing in Period 1.

Period 1: To exclude subjects with very low or very high sensitivity to tyramine, oral tyramine pressor tests will be performed prior to randomization on all subjects after eligibility has been confirmed at Screening (in the absence of any other investigational product [IP] treatment) to determine the pressor response to tyramine. The pressor response, referred to hereafter as Tyr30, is defined as the tyramine dose required to increase systolic blood pressure (SBP) by at least 30 mm Hg from daily defined baseline in three consecutive measurements within 4 hours after tyramine dosing. The test consists of daily administration of escalating doses of tyramine (up to 10 days) until a sustained SBP increase of ≥ 30 mm Hg is observed relative to the daily-defined baseline values. Sustained increase is determined by 3 consecutive SBP measurements within 4 hours after tyramine administration. The daily-defined baseline SBP value is defined as the average of five SBP measurements with approximately 5-minute interval after an initial 10- minute rest in the supine position and within 30 minutes prior to tyramine administration. Only subjects who present Tyr30 ≥ 200 mg and ≤ 800 mg will then be randomized.

Subjects will be randomized into one of three treatment groups (phenelzine, ozanimod, or placebo) in a 1:1:1 fashion while stratifying for sex in such a manner that each treatment will have a minimum of 30% of either sex.

Period 2: Subjects will receive IPs (active and/or placebo) twice daily (BID) depending on the randomization. Subjects randomized to the phenelzine group will receive phenelzine 15 mg BID for 7 days from Days 32 to 38. Subjects randomized to the ozanimod group will receive ozanimod 1.84 mg once daily (QD) for 28 days (including the initial 10-day dose escalation).

Subjects randomized to the placebo group will receive placebos for 28 days. Placebos will be matched to phenelzine or ozanimod in appearance to blind the study.

Period 3: Upon completion of Period 2, subjects in all three treatment groups will undergo a second Tyr30 test for up to 11 days. Tyramine challenge in Period 3 will remain blinded since phenelzine group has different tyramine dose schedules.

Study Population The study will enroll approximately 92 healthy men and non-pregnant, non-lactating women, ages 25 to 55 years, inclusive, with a body weight of at least 110 pounds (50 kg) and body mass index within the range of 18.0 to 30.0 kg/m2, inclusive. This is to ensure a total of 69 subjects with Tyr30 ≥ 200 mg and ≤ 800 mg at the end of Period 1 to be randomized and to allow approximately 54 subjects (18 subjects per group) to complete all three periods. A minimum of 30% of each sex will be randomized into each treatment group.

Length of Study The study duration is up to 84 ± 2 days (including a 28-day Screening period, Period 1 of up to 10 days, Period 2 of 28 days, Period 3 of up to 11 days, and a follow-up period up through 7 ± 2 days after the last dose of IP).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or non-pregnant, non-lactating woman, ages 25 to 55 years, inclusive. 2. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -1 (WOCBP only).
   * Postmenopausal (defined as 2 years after the last period and follicle-stimulating hormone (FSH) > 40 IU/L).
   * Received surgical sterilization (eg, bilateral tubal ligation, bilateral oophorectomy, hysterectomy) at least 6 months before Screening.

3. Females of child-bearing potential: Must agree to practice a highly effective method of contraception throughout the study until completion of the 75-day Safety Follow-up. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

Acceptable methods of birth control in this study are the following:

* Combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable
* Placement of an intrauterine device or intrauterine hormone-releasing system
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence

Male subjects:

Must agree to use a latex condom with spermicide during sexual contact with WOCBP while participating in the study until completion of the 75-day Safety Follow-up.

All subjects:

Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together.

4. Male subjects must agree to refrain from donating sperm during the study until 75 days after the last dose of IP.

5. Subject has a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive (Screening and Day -1 only).

6. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.

7. Subject has a mean SBP of 90 to 140 mm Hg, a DBP of 50 to 90 mm Hg from three consecutive measurements at Screening and Day -1.

8. Subject must be able to comprehend and provide written informed consent, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Subject has an unstable SBP (ie, SBP exceeds a maximum range of 10 mmHg between the lowest and highest values in three consecutive measurements within 15 minutes during Screening).
2. Subject has a presence or history of any abnormality or illness (such as glaucoma, liver disease or abnormal liver function tests) that, in the opinion of the investigator, may affect absorption, distribution, metabolism, or elimination of the IP(s) or would limit the subject's ability to participate in and complete this clinical study.
3. Subject has a history of bipolar, depression or suicidal ideation or behavior, or a history of psychiatric illnesses.
4. Subject has a history of clinically significant or unstable vascular disease, a history of syncope associated with hypotension within the last 2 years, a history of orthostatic hypotension (or SBP decrease of ≥ 20 mm Hg 2 minutes after standing compared with supine SBP), or a history of tachycardia or hypertension.
5. Subject with a seated pulse rate outside 55 to 90 bpm at Screening or Day -1.
6. Subject with a resting QTcF > 450 msec (males) or > 470 msec (females) or PR > 200 msec at Screening or Day -1.
7. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
8. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
9. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to the first dose of IP.
10. Subject has consumed any marijuana products within 3 months prior to the first dose of IP.
11. Subject has a positive urine drug test including cotinine at Screening or Day -1.
12. Subject has a positive alcohol breath test at Screening or Day -1.
13. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
14. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (including vitamins/multi-vitamins) within 14 days prior to the first dose of IP(s). St. John's wort must be discontinued at least 28 days prior to the first dose of IP.
15. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
16. Subject has used any MAO inhibitors within 90 days prior to the first dose of IP and the use of fluoxetine within 5 weeks prior to the first dose of IP.
17. Subject has a history of adverse reactions to tyramine-containing foods
18. Subject has a history of allergic reaction to tyramine, phenelzine or S1P agonist.
19. Subject has ingested alcohol within 7 days prior to the first dose of IP.
20. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
21. Subject has poor peripheral venous access.
22. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
23. Subject has a history of any medical condition or medical history that, in the opinion of the investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular | Up to approximately day 49
  Tyramine sensitivity factor (TSF) is the ratio of Tyr30 in Period 1 over Tyr30 in Period 3. Tyr30 is defined as the tyramine dose required to increase systolic blood pressure (SBP) by at least 30 mm Hg from daily defined baseline in three consecutive measurements within 4 hours after tyramine dosing.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmin | From day 11 to day 49
  Minimum observed plasma concentration within the dosing interval (Cmin)
Pharmacokinetics - Tmax | From day 11 to day 38
  Time to Cmax
Pharmacokinetics - AUC0-24 | From day 11 to day 38
  Area under the concentration-time curve from time 0 to 24 hours (AUC0-24)
Pharmacokinetics - Ctrough | From day 11 to day 49
  Pre- dose or trough concentration
Adverse Events (AEs) | From enrollment until 7 +/- 2 days after ozanimod dosing
  Number of participants with Adverse Event.
Cardiovascular Analysis-SBP | Up to approximately day 49
  Descriptive summary of systolic blood pressure by period, treatment, day and nominal time (where appropriate)
Cardiovascular Analysis-DBP | Up to approximately day 49
  Descriptive summary of diastolic blood pressure (DBP) by period, treatment, day and nominal time (where appropriate)
Cardiovascular Analysis-Heart rate | Up to approximately day 49
  Descriptive summary of heart rate by period, treatment, day and nominal time (where appropriate)
Pharmacokinetics - Cmax | From day 11 to day 38
  Maximum observed plasma concentration within the dosing interval (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States